CLINICAL TRIAL: NCT03886688
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, Dose-escalation, Pharmacokinetic Study of Single and Multiple Oral Dosing of HEC53856, A Novel HIF-PHD Inhibitor, in Healthy Non-elderly Volunteers.
Brief Title: HEC53856 Phase 1 Study - Single and Multiple Oral Dosing in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC53856-P-01
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- single ascending (Experimental): Drug or placebo, oral, fast, single dose ascending
  Interventions: Drug: HEC53856; Drug: placebo
- multiple ascending (Experimental): Drug or placebo, oral, fast, multiple dose ascending
  Interventions: Drug: HEC53856; Drug: placebo
- Food Effect (Experimental): Drug or placebo, oral, fed or fast, single dose
  Interventions: Drug: HEC53856; Drug: placebo

INTERVENTIONS:
Drug: HEC53856 — oral administration
  Other Names: HEC53856 capsule
Drug: placebo — oral administration
  Other Names: HEC53856 matching placebo capsule

SUMMARY:
To evaluate the safety, tolerability and pharmacokinetics of HEC53856 after single or multiple oral administration, as well as the food effect on the pharmacokinetics, in healthy non-elderly subjects.

DETAILED DESCRIPTION:
This is a Phase I, Single Center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Tolerability and Pharmacokinetics of HEC53856 capsule in Healthy Adult Subjects. The study consists of three parts, single dose ascending, multiple dose ascending and food effect testing. Within each part participants will be randomized to either drug or placebo.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* age: 18-45 years old(18 and 45 included).
* B.W. male> 50kg, female> 45kg, BMI - 18-28 kg/m^2
* females must not be pregnant and males and females must agree to use contraception during the study.
* able to give informed consent and comply with protocol.
* physical examination and vital signs without clinically significant abnormalities.
* agree to use contraceptive methods after informed consent acquisition through 6 months after the last administration of the study drug.

Exclusion Criteria:

* history or presence of severe gastrointestinal or systemic disorders (e.g. respiratory, endocrine, immunological, dermatological, neurological, psychiatric, renal, hepatic disease etc.)
* history or presence of significant alcoholism or drug abuse within past 5 years
* smokers, who smoke more than 5 cigarettes per day within past 3 months
* heavy drinker, namely alcohol consumption are 14 units per week (1 unit = 285 mL of beer, or 25 mL of strong wine, or 100 mL of grape wine);
* donated blood or massive blood loss within 3 months before screening (>450 mL）
* have any disease that increases the risk of bleeding or thrombus, such as acute gastritis or stomach and duodenal ulcers;
* clinically significant laboratory findings during screening
* history or presence of clinically significant ECG abnormalities
* participated in drug research study within past 3 months
* used over-the-counter/ prescription/ herbal medications/ supplements within past 14 days.
* Strenuous activity (as assessed by the investigator) is prohibited from 2 weeks prior to admission until discharge from the unit.
* female in pregnancy or lactation.
* viral hepatitis（including CHB and CHC）and positive test result of anti-HIV Ab or syphilis.
* the investigator believes that the one should not be included

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events [Safety and Tolerability] | Up to Day 10 after last dose
  To assess the safety and tolerability by incidence of treatment-emergent adverse events after a single dose or multiple doses of HEC53856 capsule

SECONDARY OUTCOMES:
AUC0-t | Up to 96 hours after dosing
  Area under the concentration versus time curve (AUC) from time zero to the time of the last quantifiable concentration
Cmax | Up to 96 hours after dosing
  Maximum observed plasma concentration
Tmax | Up to 96 hours after dosing
  Time of the maximum observed plasma concentration
T T½ | Up to 96 hours after dosing
  Apparent terminal elimination half-life

OTHER OUTCOMES:
Vz/F | Up to 96 hours after dosing
  Apparent volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Ding Yanhua, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China